CLINICAL TRIAL: NCT03689374
Title: Effect of Semaglutide Once-weekly Versus Insulin Aspart Three Times Daily, Both as Add on to Metformin and Optimised Insulin Glargine (U100) in Subjects With Type 2 Diabetes A 52-week, Multi-centre, Multinational, Open-label, Active-controlled, Two Armed, Parallel-group, Randomised Trial in Subjects With Type 2 Diabetes
Brief Title: A Research Study to Compare Semaglutide to Insulin Aspart, When Taken Together With Metformin and Insulin Glargine, in People With Type 2 Diabetes
Acronym: SUSTAIN 11
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9535-4386; U1111-1200-0164 (Other: World Health Organization (WHO)); 2017-003219-20 (Registry Identifier: EudraCT)
Record Dates: First submitted 2018-09-27; First posted 2018-09-28 (Actual); Results first posted 2022-05-04 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Semaglutide (Experimental): Run-in period (12 weeks): subjects will be treated with metformin and insulin glargine (IGlar) U100.
  Treatment period: Participants who are not in glycaemic control (defined as HbA1c of more than or equal to 7.5% to less than or equal to 10%) after run-in will receive semaglutide for 52 weeks in addition to metformin and IGlar U100.
  Metformin will be considered as background therapy during the trial.
  Interventions: Drug: Semaglutide; Drug: Insulin glargine U100
- Insulin aspart (Active Comparator): Run-in period (12 weeks): subjects will be treated with metformin and insulin IGlar U100.
  Treatment period: Participants who are not in glycaemic control (defined as HbA1c of more than or equal to 7.5% to less than or equal to 10%) after run-in receive insulin aspart for 52 weeks in addition to metformin and IGlar U100.
  Metformin will be considered as background therapy during the trial.
  Interventions: Drug: Insulin aspart; Drug: Insulin glargine U100

INTERVENTIONS:
Drug: Semaglutide — Subjects will receive subcutaneous (s.c., under the skin) injections of semaglutide once weekly (OW) with a dose of 0.25 mg. The dose should be increased after four weeks to 0.5 mg semaglutide. After 4 more weeks the dose can be increased to 1.0 mg semaglutide if the study doctor decides and further dose adjusted throughout the study.
  Arms: Semaglutide
Drug: Insulin aspart — Subjects should initiate treatment with 4U of Insulin aspart (s.c. injections) before each main meal, three times daily (TID). The dose will be adjusted individually based on pre-prandial and bedtime self measured plasma glucose (SMPG) from the preceding 3 days
  Arms: Insulin aspart
Drug: Insulin glargine U100 — Run-in period: Subjects will receive s.c. injections of IGlar U100 OD in accordance with the approved local label of IGlar U100. The dose will be adjusted based on the mean of three pre-breakfast SMPG values (target SMPG: 4.0-6.9 mmol/L)

SUMMARY:
This study will compare the effect of semaglutide once weekly to insulin aspart 3 times daily as add on to metformin and insulin glargine in people with type 2 diabetes. Participants will either get insulin glargine and semaglutide or insulin glargine and insulin aspart - which treatment the participant get is decided by chance. Insulin glargine is taken once a day and semaglutide once a week. Insulin aspart is taken three times per day before a meal. All three medicines come in pre-filled pens for injection under the skin. The study will last for about 71 weeks. If participant's blood sugar gets under or over certain values participant will only participate in 14 weeks. The study doctor will inform the participant about this. The participant will have 15 clinic visits and 22 phone calls with the study doctor.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age greater than or equal to 18 years at the time of signing informed consent
* Diagnosed with type 2 diabetes greater than or equal to 180 days prior to the day of screening
* Treated with basal insulin once daily or twice daily for greater than or equal to 90 days prior to the day of screening
* Stable daily dose for 90 days prior to the day of screening of the following anti-diabetic drugs or combination regimens: Any metformin formulations (greater than or equal to 1500 mg to less than or equal to 3000 mg or maximum tolerated or effective dose documented in subject's medical record), alone or in combination (including fixed-dose drug combination) with up to one additional of the following oral antidiabetic drugs: sulfonylureas, meglitinides, dipeptidyl peptidase-4 inhibitors or alpha-glucosidase inhibitors
* Glycated haemoglobin (HbA1c) of greater than 7.5% to less than or less than or equal to 10.0% (greater than 58 mmol/mol to less than or equal to 86 mmol/mol)

Exclusion Criteria:

* History or presence of pancreatitis (acute or chronic)
* Any of the following: myocardial infarction, stroke, hospitalization for unstable angina or transient ischaemic attack within the past 180 days prior to the day of screening
* Subjects presently classified as being in New York Heart Association Class IV
* Planned coronary, carotid or peripheral artery revascularisation known on the day of screening
* Treatment with any medication for the indication of diabetes or obesity other than stated in the inclusion criteria within the past 90 days prior to the day of screening. However, short term bolus insulin treatment for a maximum of 14 days prior to the day of screening is allowed
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a pharmacologically pupil-dilated fundus examination performed by an ophthalmologist or an equally qualified health care provider (for example, optometrist) within the past 90 days prior to run-in

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2274 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2021-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (160):
- Bosnia and Herzegovina (3):
  - Novo Nordisk Investigational Site, Banja Luka
  - Novo Nordisk Investigational Site, Sarajevo
  - Novo Nordisk Investigational Site, Tuzla
- Bulgaria (8):
  - Novo Nordisk Investigational Site, Burgas
  - Novo Nordisk Investigational Site, Byala
  - Novo Nordisk Investigational Site, Dimitrovgrad
  - Novo Nordisk Investigational Site, Plovdiv
  - Novo Nordisk Investigational Site, Rousse
  - Novo Nordisk Investigational Site, Sofia
  - Novo Nordisk Investigational Site, Stara Zagora
  - Novo Nordisk Investigational Site, Varna
- Croatia (6):
  - Novo Nordisk Investigational Site, Karlovac
  - Novo Nordisk Investigational Site, Osijek
  - Novo Nordisk Investigational Site, Pula
  - Novo Nordisk Investigational Site, Rijeka
  - Novo Nordisk Investigational Site, Varaždin
  - Novo Nordisk Investigational Site, Zagreb
- Czechia (8):
  - Novo Nordisk Investigational Site, Beroun
  - Novo Nordisk Investigational Site, Brno
  - Novo Nordisk Investigational Site, Kladno - Krocehlavy
  - Novo Nordisk Investigational Site, Mladá Boleslav
  - Novo Nordisk Investigational Site, Náchod
  - Novo Nordisk Investigational Site, Olomouc
  - Novo Nordisk Investigational Site, Pilsen
  - Novo Nordisk Investigational Site, Prostějov
- Estonia (3):
  - Novo Nordisk Investigational Site, Pärnu
  - Novo Nordisk Investigational Site, Tallinn
  - Novo Nordisk Investigational Site, Viljandi
- Germany (23):
  - Novo Nordisk Investigational Site, Bad Kreuznach
  - Novo Nordisk Investigational Site, Bad Mergentheim
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Eisenach
  - Novo Nordisk Investigational Site, Essen
  - Novo Nordisk Investigational Site, Esslingen am Neckar
  - Novo Nordisk Investigational Site, Falkensee
  - Novo Nordisk Investigational Site, Friedrichsthal
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Hohenmölsen
  - Novo Nordisk Investigational Site, Jerichow
  - Novo Nordisk Investigational Site, Kiel Kronshagen
  - Novo Nordisk Investigational Site, Leipzig
  - Novo Nordisk Investigational Site, Münster
  - Novo Nordisk Investigational Site, Oldenburg I. Holst
  - Novo Nordisk Investigational Site, Pohlheim
  - Novo Nordisk Investigational Site, Rehlingen-Siersburg
  - Novo Nordisk Investigational Site, Saint Ingbert-Oberwürzbach
  - Novo Nordisk Investigational Site, Schwabenheim
  - Novo Nordisk Investigational Site, Schweinfurt
  - Novo Nordisk Investigational Site, Stuhr
  - Novo Nordisk Investigational Site, Stuttgart
  - Novo Nordisk Investigational Site, Villingen-Schwenningen
- Greece (5):
  - Novo Nordisk Investigational Site, Alexandroupoli
  - Novo Nordisk Investigational Site, Athens
  - Novo Nordisk Investigational Site, Larissa
  - Novo Nordisk Investigational Site, Piraeus
  - Novo Nordisk Investigational Site, Thessaloniki
- Hungary (7):
  - Novo Nordisk Investigational Site, Budapest
  - Novo Nordisk Investigational Site, Gyula
  - Novo Nordisk Investigational Site, Nagykanizsa
  - Novo Nordisk Investigational Site, Pécs
  - Novo Nordisk Investigational Site, Salgótarján
  - Novo Nordisk Investigational Site, Szeged
  - Novo Nordisk Investigational Site, Zalaegerszeg
- India (19):
  - Novo Nordisk Investigational Site, Hyderabad, Andhra Pradesh
  - Novo Nordisk Investigational Site, Ahmedabad, Gujarat
  - Novo Nordisk Investigational Site, Bangalore, Karnataka
  - Novo Nordisk Investigational Site, Indore, Madhya Pradesh
  - Novo Nordisk Investigational Site, Mumbai, Maharashtra
  - Novo Nordisk Investigational Site, Nagpur, Maharashtra
  - Novo Nordisk Investigational Site, Pune, Maharashtra
  - Novo Nordisk Investigational Site, Delhi, New Delhi
  - Novo Nordisk Investigational Site, New Dehli, New Delhi
  - Novo Nordisk Investigational Site, Bhubaneswar, Odisha
  - Novo Nordisk Investigational Site, Chandigarh, Punjab
  - Novo Nordisk Investigational Site, Ludhiana, Punjab
  - Novo Nordisk Investigational Site, Mohali, Punjab
  - Novo Nordisk Investigational Site, Jaipur, Rajasthan
  - Novo Nordisk Investigational Site, Madurai, Tamil Nadu
  - Novo Nordisk Investigational Site, Hyderabad, Telangana
  - Novo Nordisk Investigational Site, Hyderbad, Telangana
  - Novo Nordisk Investigational Site, Kolkata, West Bengal
  - Novo Nordisk Investigational Site, New Delhi
- Latvia (5):
  - Novo Nordisk Investigational Site, Jelgava
  - Novo Nordisk Investigational Site, Ogre
  - Novo Nordisk Investigational Site, Riga
  - Novo Nordisk Investigational Site, Sigulda
  - Novo Nordisk Investigational Site, Talsi
- Lithuania (3):
  - Novo Nordisk Investigational Site, Kaunas
  - Novo Nordisk Investigational Site, Panevezys
  - Novo Nordisk Investigational Site, Vilnius
- Novo Nordisk Investigational Site, Skopje, North Macedonia
- Poland (13):
  - Novo Nordisk Investigational Site, Bialystok
  - Novo Nordisk Investigational Site, Gorzów Wielkopolski
  - Novo Nordisk Investigational Site, Lodz
  - Novo Nordisk Investigational Site, Lublin
  - Novo Nordisk Investigational Site, Poznan
  - Novo Nordisk Investigational Site, Puławy
  - Novo Nordisk Investigational Site, Ruda Śląska
  - Novo Nordisk Investigational Site, Siedlce
  - Novo Nordisk Investigational Site, Skorzewo
  - Novo Nordisk Investigational Site, Warsaw
  - Novo Nordisk Investigational Site, Wierzchosławice
  - Novo Nordisk Investigational Site, Wroclaw
  - Novo Nordisk Investigational Site, Zabrze
- Portugal (7):
  - Novo Nordisk Investigational Site, Almada
  - Novo Nordisk Investigational Site, Braga
  - Novo Nordisk Investigational Site, Coimbra
  - Novo Nordisk Investigational Site, Lisbon
  - Novo Nordisk Investigational Site, Loures
  - Novo Nordisk Investigational Site, Porto
  - Novo Nordisk Investigational Site, Setúbal
- Romania (6):
  - Novo Nordisk Investigational Site, Cluj-Napoca, Cluj
  - Novo Nordisk Investigational Site, Târgovişte, Dâmbovița County
  - Novo Nordisk Investigational Site, Târgu Mureş, Mureș County
  - Novo Nordisk Investigational Site, Ploieşti, Prahova
  - Novo Nordisk Investigational Site, Brasov
  - Novo Nordisk Investigational Site, Galati
- Serbia (5):
  - Novo Nordisk Investigational Site, Belgrade
  - Novo Nordisk Investigational Site, Kragujevac
  - Novo Nordisk Investigational Site, Niš
  - Novo Nordisk Investigational Site, Novi Sad
  - Novo Nordisk Investigational Site, Zaječar
- Slovakia (9):
  - Novo Nordisk Investigational Site, Bardejov
  - Novo Nordisk Investigational Site, Bratislava
  - Novo Nordisk Investigational Site, Dolný Kubín
  - Novo Nordisk Investigational Site, Levice
  - Novo Nordisk Investigational Site, Ľubochňa
  - Novo Nordisk Investigational Site, Martin
  - Novo Nordisk Investigational Site, Prešov
  - Novo Nordisk Investigational Site, Prievidza
  - Novo Nordisk Investigational Site, Sabinov
- Slovenia (5):
  - Novo Nordisk Investigational Site, Brežice
  - Novo Nordisk Investigational Site, Jesenice
  - Novo Nordisk Investigational Site, Koper
  - Novo Nordisk Investigational Site, Murska Sobota
  - Novo Nordisk Investigational Site, Nova Gorica
- South Africa (7):
  - Novo Nordisk Investigational Site, Benoni, Gauteng
  - Novo Nordisk Investigational Site, Cosmo City, Gauteng
  - Novo Nordisk Investigational Site, Johannesburg, Gauteng
  - Novo Nordisk Investigational Site, Lenasia, Gauteng
  - Novo Nordisk Investigational Site, Pretoria, Gauteng
  - Novo Nordisk Investigational Site, Durban, KwaZulu-Natal
  - Novo Nordisk Investigational Site, eMkhomazi, KwaZulu-Natal
- Spain (9):
  - Novo Nordisk Investigational Site, Almería
  - Novo Nordisk Investigational Site, Antequera
  - Novo Nordisk Investigational Site, Córdoba
  - Novo Nordisk Investigational Site, Fuenlabrada - Madrid
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, Málaga
  - Novo Nordisk Investigational Site, Palma de Mallorca
  - Novo Nordisk Investigational Site, Segovia
  - Novo Nordisk Investigational Site, Seville
- Turkey (Türkiye) (8):
  - Novo Nordisk Investigational Site, Adana
  - Novo Nordisk Investigational Site, Ankara
  - Novo Nordisk Investigational Site, Antalya
  - Novo Nordisk Investigational Site, Denizli
  - Novo Nordisk Investigational Site, Erzurum
  - Novo Nordisk Investigational Site, Istanbul
  - Novo Nordisk Investigational Site, Izmir
  - Novo Nordisk Investigational Site, Trabzon

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Result] Kellerer M, Kaltoft MS, Lawson J, Nielsen LL, Strojek K, Tabak O, Jacob S. Effect of once-weekly semaglutide versus thrice-daily insulin aspart, both as add-on to metformin and optimized insulin glargine treatment in participants with type 2 diabetes (SUSTAIN 11): A randomized, open-label, multinational, phase 3b trial. Diabetes Obes Metab. 2022 Sep;24(9):1788-1799. doi: 10.1111/dom.14765. Epub 2022 Jun 29. PMID 35546450

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 209 sites in 21 countries: Bosnia-Herzegovina (3 sites), Bulgaria (9 sites), Croatia (7 sites), Czech Republic (7 sites), Estonia (5 sites), Germany (25 sites), Greece (14 sites), Hungary (8 sites), India (20 sites), Latvia (7 sites), Lithuania (6 sites), Macedonia (3 sites), Poland (20 sites), Portugal (6 sites), Romania (7 sites), Serbia (14 sites), Slovakia (9 sites), Slovenia (6 sites), South Africa (11 sites), Spain (8 sites) and Turkey (14 sites).
Pre-assignment Details: This trial consisted of 12-week run-in, 52-week treatment period and participants were followed up 5 weeks for safety. Participants were randomized 1:1 to receive treatment with: metformin + insulin glargine (IGlar) U100 + once-weekly semaglutide subcutaneously (s.c). or metformin + insulin glargine U100 + mealtime insulin aspart s.c. three times daily.
Groups:
- All Participants: During run-in period insulin glargine in combination with metformin was to be optimized. All enrolled participants received metformin orally and IGlar U100 s.c. injection in run-in period. Metformin was optimized in dose range of greater than or equal to (>=) 1500 milligrams (mg) to less than or equal to (<=) 3000 mg. After run-in period, participants were randomized 1:1 to receive add-on treatment with semaglutide once weekly or insulin aspart three times daily (TID) in treatment period.
- Semaglutide: Participants received metformin, IGlar U100 and semaglutide for 52 weeks in treatment period. Metformin dose was maintained at same level and frequency as optimized in run-in period unless safety concern related to background medication arose; IGlar U100 dose was adjusted in run-in period, increases in IGlar U100 dose was based on mean of 3 prebreakfast self-measured plasma glucose (SMPG) values obtained on day of visit/telephone contact and 2 days before contact and dose reduction of IGlar U100 was considered in accordance with approved local label to reduce risk of hypoglycaemia. Participants self-administered s.c. injection of semaglutide at an initiation dose of 0.25 mg once weekly, after 4 weeks dose was increased to 0.5 mg, and 1 mg after at least 4 weeks to further improve glycaemic control, at investigator's discretion. Dose reduction from 1 to 0.5 mg was allowed in case of safety concern/unacceptable intolerability. Participants were followed up for 5 weeks (week 57) for safety.
- Insulin Aspart: Participants received metformin, IGlar U100 and insulin aspart for 52 weeks in treatment period. Metformin dose was maintained at same level and frequency as optimized in run-in period unless safety concern related to background medication arose; IGlar U100 dose was adjusted in run-in period, increases in IGlar U100 dose was based on mean of 3 prebreakfast SMPG values obtained on day of visit/telephone contact and 2 days before contact and dose reduction of IGlar U100 was considered in accordance with approved local label to reduce risk of hypoglycaemia. Participants self-administered s.c. injection of insulin aspart at an initiation dose of 4 units three times daily, dose adjustments were considered twice weekly based on pre-prandial and bedtime SMPG from the preceding 3 days and the individualized goal according to investigator's discretion. Participants were followed up for 5 weeks (week 57) for safety.
Period: Run-in Period (12 Weeks)
Arm/Group | All Participants | Semaglutide | Insulin Aspart
Started | 2274 | 0 | 0
Completed | 1748 | 0 | 0
Not Completed | 526 | 0 | 0
Not completed — Run-in failure | 526 | 0 | 0
Period: Treatment Period (Week 0 to 52)
Arm/Group | All Participants | Semaglutide | Insulin Aspart
Started | 0 | 874 | 874
Treated | 0 | 874 | 864
Full Analysis Set | 0 | 874 | 874
Safety Analysis Set | 0 | 874 | 864
Completed | 0 | 850 | 831
Not Completed | 0 | 24 | 43
Not completed — Withdrawal by Subject | 0 | 10 | 38
Not completed — Lost to Follow-up | 0 | 3 | 4
Not completed — Death | 0 | 11 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Semaglutide | Insulin Aspart | Total
Number analyzed (Participants) | 874 | 874 | 1748
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.8 (9.4) | 61.5 (9.5) | 61.2 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 429 | 425 | 854
  Male | 445 | 449 | 894
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 22 | 45
  Not Hispanic or Latino | 851 | 852 | 1703
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska native | 0 | 0 | 0
  Race: Asian | 176 | 166 | 342
  Race: Black or African American | 21 | 14 | 35
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Race: White | 674 | 691 | 1365
  Race: Other | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycated Haemoglobin (HbA1c)
Description: Change from baseline in HbA1c at week 52 is presented. Data is reported for 'on-treatment' observation period: from the date of first dose of trial product (week 0) to the last date on trial product with a visit window of +7 days (week 52).
Time Frame: Baseline (week 0), week 52
Population: Full analysis set included all randomized participants. Overall Number of Participants Analyzed = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Semaglutide | Insulin Aspart
Number analyzed (Participants) | 795 | 783
Percentage of HbA1c | -1.5 (1.0) | -1.2 (1.0)
Statistical Analysis 1: Comparison: Semaglutide vs Insulin Aspart; Test type: Non-Inferiority — The responses were analyzed using an ANCOVA with treatment as fixed factor and baseline value as a covariate. Before analysis, missing data were multiple imputed using observed data from participants within the same group defined by randomized treatment, using a regression model including randomized treatment group and data from baseline and all previous visits as covariates. The prespecified non inferiority margin was 0.3%-point; p < 0.0001, t-distributed test; The non-inferiority p-value was calculated as two times the one-sided p-value from a t-distributed test; Treatment difference = -0.29, 95% CI 2-sided [-0.38 to -0.20]

2. Secondary Outcome: Time to First Event Adjudication Committee (EAC)-Confirmed Severe Hypoglycaemic Episode American Diabetes Association (ADA) From Randomization up to Week 52
Description: First event per 100 years of exposure time for first EAC confirmed severe hypoglycaemic episodes from randomization (week 0) to week 52 are presented. As per 2013 ADA criteria severe hypoglycaemic episodes were episodes with plasma glucose (PG) less than or equal to (<=) 3.9 millimoles per liter (mmol/L) (70 milligrams per deciliter (mg/dL)). EAC confirmed-severe hypoglycaemia was an episode requiring assistance of another person to actively administer carbohydrate, glucagon or take other corrective actions. Data is reported for 'on-treatment' observation period: from the date of first dose of trial product (week 0) to the last date on trial product with a visit window of +7 days (week 52).
Time Frame: From randomization (week 0) up to week 52
Population: as for outcome 1
Measure: Number; unit: First event per 100 years of exposure
Arm/Group | Semaglutide | Insulin Aspart
Number analyzed (Participants) | 874 | 864
First event per 100 years of exposure | 0.4 | 0.7

3. Secondary Outcome: Time to First Event Adjudication Committee-confirmed Severe Hypoglycaemic Episode (ADA) Requiring Hospitalization, Documented Medical Help, or is Life-threatening Randomization up to Week 52
Description: First event per 100 years of exposure time for first EAC confirmed severe hypoglycaemic episodes requiring hospitalization, documented medical help, or is life threatening from randomization (week 0) to week 52 are presented. As per 2013 ADA criteria severe hypoglycaemic episodes were episodes with PG <=3.9 mmol/L (70 mg/dL). EAC confirmed-severe hypoglycaemia was an episode requiring assistance of another person to actively administer carbohydrate, glucagon or take other corrective actions. Data is reported for 'on-treatment' observation period: from the date of first dose of trial product (week 0) to the last date on trial product with a visit window of +7 days (week 52).
Time Frame: From randomization (week 0) up to week 52
Population: as for outcome 1
Measure: Number; unit: First event per 100 years of exposure
Arm/Group | Semaglutide | Insulin Aspart
Number analyzed (Participants) | 874 | 864
First event per 100 years of exposure | 0.2 | 0.4

4. Secondary Outcome: Number of Event Adjudication Committee-confirmed Severe Hypoglycaemic Episodes (ADA) From Randomization to Week 52
Description: Number of EAC-confirmed severe hypoglycaemic episodes from randomization (week 0) up to week 52 are presented. As per 2013 ADA criteria severe hypoglycaemic episodes were episodes with PG <=3.9 mmol/L (70 mg/dL). EAC confirmed-severe hypoglycaemia was an episode requiring assistance of another person to actively administer carbohydrate, glucagon or take other corrective actions. Data is reported for 'on-treatment' observation period: from the date of first dose of trial product (week 0) to the last date on trial product with a visit window of +7 days (week 52).
Time Frame: From randomization (week 0) to week 52
Population: Full analysis set included all randomized participants.
Measure: Number; unit: Episodes
Arm/Group | Semaglutide | Insulin Aspart
Number analyzed (Participants) | 874 | 874
Episodes | 4 | 7

5. Secondary Outcome: Number of Event Adjudication Committee-confirmed Severe (ADA) or Blood Glucose (BG) Confirmed, Symptomatic Hypoglycaemic Episodes (Plasma Glucose Less Than (<) 3.1 mmol/L (56 mg/dL)) From Randomization to Week 52
Description: Number of EAC-confirmed severe or BG confirmed, symptomatic hypoglycaemic episodes (PG <3.1 mmol/L (56 mg/dL)) from randomization (week 0) to week 52 are presented. As per 2013 ADA criteria severe hypoglycaemic episodes were episodes with PG <=3.9 mmol/L (70 mg/dL). Severe or BG confirmed symptomatic hypoglycaemia was an episode, that was BG confirmed by PG value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia. Data is reported for 'on-treatment' observation period: from the date of first dose of trial product (week 0) to the last date on trial product with a visit window of +7 days (week 52).
Time Frame: From randomization (week 0) to week 52
Population: Full analysis set included all randomized participants.
Measure: Number; unit: Episodes
Arm/Group | Semaglutide | Insulin Aspart
Number analyzed (Participants) | 874 | 874
Episodes | 254 | 1744

6. Secondary Outcome: Number of Event Adjudication Committee-confirmed Severe (ADA) or Blood Glucose Confirmed, Symptomatic Hypoglycaemic Episodes (Plasma Glucose <= 3.9 mmol/L (70 mg/dL)) From Randomization to Week 52
Description: Number of EAC-confirmed severe or BG confirmed, symptomatic hypoglycaemic episodes (PG <=3.9 mmol/L (70 mg/dL)) from randomization (week 0) to week 52 are presented. As per 2013 ADA criteria severe hypoglycaemic episodes were episodes with PG <=3.9 mmol/L (70 mg/dL). Severe or BG confirmed symptomatic hypoglycaemia was an episode during which symptoms of hypoglycaemia were not accompanied by a PG determination but that was presumably caused by a PG concentration <= 3.9 mmol/L (70 mg/dL). Data is reported for 'on-treatment' observation period: from the date of first dose of trial product (week 0) to the last date on trial product with a visit window of +7 days (week 52).
Time Frame: From randomization (week 0) to week 52
Population: Full analysis set included all randomized participants.
Measure: Number; unit: Episodes
Arm/Group | Semaglutide | Insulin Aspart
Number analyzed (Participants) | 874 | 874
Episodes | 1420 | 5616

7. Secondary Outcome: Number of Event Adjudication Committee-confirmed Severe Hypoglycaemic Episodes (ADA) Requiring Hospitalization, Documented Medical Help, or is Life-threatening From Randomization to Week 52
Description: Number of EAC-confirmed severe hypoglycaemic episodes requiring hospitalization, documented medical help, or is life-threatening from randomization (week 0) to week 52 are presented. As per 2013 ADA criteria severe hypoglycaemic episodes were episodes with PG <=3.9 mmol/L (70 mg/dL). Severe hypoglycaemia was an episode requiring assistance of another person to actively administer carbohydrate, glucagon or take other corrective actions. Data is reported for 'on-treatment' observation period: from the date of first dose of trial product (week 0) to the last date on trial product with a visit window of +7 days (week 52).
Time Frame: From randomization (week 0) to week 52
Population: Full analysis set included all randomized participants.
Measure: Number; unit: Episodes
Arm/Group | Semaglutide | Insulin Aspart
Number analyzed (Participants) | 874 | 874
Episodes | 2 | 4

8. Secondary Outcome: Number of Event Adjudication Committee-confirmed Severe (ADA) or Clinically Significant Hypoglycaemic Episodes (Plasma Glucose < 3.0 mmol/L (54 mg/dL)) From Randomization to Week 52
Description: Number of EAC-confirmed severe or clinically significant hypoglycaemic episodes (plasma glucose < 3.0 mmol/L (54 mg/dL)) from randomization (week 0) to week 52 are presented. As per 2013 ADA criteria severe hypoglycaemic episodes were episodes with PG <=3.9 mmol/L (70 mg/dL). Severe hypoglycaemia was an episode requiring assistance of another person to actively administer carbohydrate, glucagon or take other corrective actions. Hypoglycaemic episode with plasma glucose < 3.0 mmol/L (54 mg/dL)) was considered as clinically significant. Data is reported for 'on-treatment' observation period: from the date of first dose of trial product (week 0) to the last date on trial product with a visit window of +7 days (week 52).
Time Frame: From randomization (week 0) to week 52
Population: Full analysis set included all randomized participants.
Measure: Number; unit: Episodes
Arm/Group | Semaglutide | Insulin Aspart
Number analyzed (Participants) | 874 | 874
Episodes | 339 | 2270

9. Secondary Outcome: Daily Basal Insulin Dose at Week 52
Description: Daily basal insulin dose at week 52 is presented. Data is reported for 'on-treatment' observation period: from the date of first dose of trial product (week 0) to the last date on trial product with a visit window of +7 days (week 52).
Time Frame: At week 52
Population: Safety analysis set included all participants exposed to at least one dose of trial product. Overall Number of Participants Analyzed = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units of insulin
Arm/Group | Semaglutide | Insulin Aspart
Number analyzed (Participants) | 803 | 794
Units of insulin | 35.8 (19.4) | 40.7 (22.0)

10. Secondary Outcome: Total Daily Insulin Dose at Week 52
Description: Total daily insulin dose at week 52 is presented. Data is reported for 'on-treatment' observation period: from the date of first dose of trial product (week 0) to the last date on trial product with a visit window of +7 days (week 52).
Time Frame: At week 52
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units of insulin
Arm/Group | Semaglutide | Insulin Aspart
Number analyzed (Participants) | 803 | 797
Units of insulin | 35.8 (19.4) | 77.7 (40.0)

11. Secondary Outcome: Change From Baseline to Week 52 in Body Weight (Kilogram (kg))
Description: Change from baseline in body weight at week 52 is presented. Data is reported for 'on-treatment' observation period: from the date of first dose of trial product (week 0) to the last date on trial product with a visit window of +7 days (week 52).
Time Frame: Baseline (week 0), week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Semaglutide | Insulin Aspart
Number analyzed (Participants) | 801 | 793
kilograms | -4.2 (4.6) | 2.9 (4.1)

12. Secondary Outcome: Change From Baseline to Week 52 in Fasting Plasma Glucose (FPG)
Description: Change from baseline in FPG at week 52 is presented. Data is reported for 'on-treatment' observation period: from the date of first dose of trial product (week 0) to the last date on trial product with a visit window of +7 days (week 52).
Time Frame: Baseline (week 0), week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | Semaglutide | Insulin Aspart
Number analyzed (Participants) | 770 | 762
millimoles per liter (mmol/L) | -1.3 (2.9) | -0.8 (3.1)

13. Secondary Outcome: Change From Baseline to Week 52 in 7-point Self-measured Plasma Glucose Profile (SMPG ): Mean 7-point Profile (7-PP)
Description: Change from baseline in 7-point self-measured plasma glucose profile: mean 7-PP at week 52 is presented. All participants were instructed to perform 7-point SMPG profiles before breakfast, 90 minutes after the start of breakfast, before lunch, 90 minutes after the start of lunch, before main evening meal (dinner), 90 minutes after the start of main evening meal (dinner) and at bedtime. The measurements were to be performed before any injection of bolus insulin and just before the start of the meal (breakfast, lunch or main evening meal), and values measured before breakfast were performed in a fasting condition. Data is reported for 'on-treatment' observation period: from the date of first dose of trial product (week 0) to the last date on trial product with a visit window of +7 days (week 52).
Time Frame: Baseline (week 0), week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Semaglutide | Insulin Aspart
Number analyzed (Participants) | 757 | 737
mmol/L | -2.1 (2.0) | -2.1 (2.0)

14. Secondary Outcome: Change From Baseline to Week 52 in 7-point Self-measured Plasma Glucose Profile: Mean Post-prandial Increment (Over All Meals)
Description: Change from baseline in 7-point SMPG profile: mean post-prandial increment (over all meals) at week 52 is presented. Data is reported for 'on-treatment' observation period: from the date of first dose of trial product (week 0) to the last date on trial product with a visit window of +7 days (week 52).
Time Frame: Baseline (week 0), week 52
Population: Full analysis set included all randomized participants. Overall Number of Participants Analyzed = participants with available data for this outcome measure .
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Semaglutide | Insulin Aspart
Number analyzed (Participants) | 747 | 724
mmol/L | -0.7 (1.8) | -0.9 (2.1)

15. Secondary Outcome: Change From Baseline to Week 52 in Body Mass Index (BMI)
Description: Change from baseline in BMI at week 52 is presented. Data is reported for 'on-treatment' observation period: from the date of first dose of trial product (week 0) to the last date on trial product with a visit window of +7 days (week 52).
Time Frame: Baseline (week 0), week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kilograms per meter square (kg/m^2)
Arm/Group | Semaglutide | Insulin Aspart
Number analyzed (Participants) | 801 | 793
kilograms per meter square (kg/m^2) | -1.5 (1.7) | 1.0 (1.5)

16. Secondary Outcome: Change From Baseline to Week 52 in Waist Circumference
Description: Change from baseline in waist circumference at week 52 is presented. Data is reported for 'on-treatment' observation period: from the date of first dose of trial product (week 0) to the last date on trial product with a visit window of +7 days (week 52).
Time Frame: Baseline (week 0), week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: centimeters (cm)
Arm/Group | Semaglutide | Insulin Aspart
Number analyzed (Participants) | 799 | 793
centimeters (cm) | -3.3 (5.6) | 2.1 (4.9)

17. Secondary Outcome: Change From Baseline to Week 52 in Body Weight (Percentage): Ratio to Baseline
Description: Change from baseline in body weight (measured in percentage) at week 52 is presented as ratio to baseline. Data is reported for 'on-treatment' observation period: from the date of first dose of trial product (week 0) to the last date on trial product with a visit window of +7 days (week 52).
Time Frame: Baseline (week 0), week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio of body weight
Arm/Group | Semaglutide | Insulin Aspart
Number analyzed (Participants) | 801 | 793
Ratio of body weight | 1.0 (0.1) | 1.0 (0.0)

18. Secondary Outcome: Change From Baseline to Week 52 in Fasting Blood Lipids: Total Cholesterol (Ratio to Baseline)
Description: Change from baseline in total cholesterol (measured in mmol/L) at week 52 is presented as ratio to baseline. Data is reported for 'on-treatment' observation period: from the date of first dose of trial product (week 0) to the last date on trial product with a visit window of +7 days (week 52).
Time Frame: Baseline (week 0), week 52
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of total cholesterol
Arm/Group | Semaglutide | Insulin Aspart
Number analyzed (Participants) | 792 | 784
Ratio of total cholesterol | 1.0 (19.6) | 1.0 (20.9)

19. Secondary Outcome: Change From Baseline to Week 52 in Fasting Blood Lipids: Low-density Lipoprotein (LDL) Cholesterol (Ratio to Baseline)
Description: Change from baseline in LDL cholesterol (measured in mmol/L) at week 52 is presented as ratio to baseline. Data is reported for 'on-treatment' observation period: from the date of first dose of trial product (week 0) to the last date on trial product with a visit window of +7 days (week 52).
Time Frame: Baseline (week 0), week 52
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of LDL cholesterol
Arm/Group | Semaglutide | Insulin Aspart
Number analyzed (Participants) | 789 | 781
Ratio of LDL cholesterol | 1.0 (36.2) | 1.0 (35.2)

20. Secondary Outcome: Change From Baseline to Week 52 in Fasting Blood Lipids: High-density Lipoprotein (HDL) Cholesterol (Ratio to Baseline)
Description: Change from baseline in HDL cholesterol (measured in mmol/L) at week 52 is presented as ratio to baseline. Data is reported for 'on-treatment' observation period: from the date of first dose of trial product (week 0) to the last date on trial product with a visit window of +7 days (week 52).
Time Frame: Baseline (week 0), week 52
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of HDL cholesterol
Arm/Group | Semaglutide | Insulin Aspart
Number analyzed (Participants) | 751 | 741
Ratio of HDL cholesterol | 1.0 (16.7) | 1.0 (16.4)

21. Secondary Outcome: Change From Baseline to Week 52 in Fasting Blood Lipids: Triglycerides (Ratio to Baseline)
Description: Change from baseline in triglycerides (measured in mmol/L) at week 52 is presented as ratio to baseline. Data is reported for 'on-treatment' observation period: from the date of first dose of trial product (week 0) to the last date on trial product with a visit window of +7 days (week 52).
Time Frame: Baseline (week 0), week 52
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of triglycerides
Arm/Group | Semaglutide | Insulin Aspart
Number analyzed (Participants) | 789 | 781
Ratio of triglycerides | 0.9 (40.4) | 1.0 (42.0)

22. Secondary Outcome: Change From Baseline to Week 52 in Systolic and Diastolic Blood Pressure
Description: Change from baseline in systolic and diastolic blood pressure at week 52 are presented. Data is reported for 'on-treatment' observation period: from the date of first dose of trial product (week 0) to the last date on trial product with a visit window of +7 days (week 52).
Time Frame: Baseline (week 0), week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Semaglutide | Insulin Aspart
Number analyzed (Participants) | 784 | 765
millimeter of mercury (mmHg)
  Diastolic Blood Pressure | -1.4 (8.7) | -0.4 (9.0)
  Systolic Blood Pressure | -2.8 (13.8) | 1.0 (14.0)

23. Secondary Outcome: Change From Baseline to Week 52 in Pulse Rate
Description: Change from baseline in pulse rate at week 52 is presented. Data is reported for 'on-treatment' observation period: from the date of first dose of trial product (week 0) to the last date on trial product with a visit window of +7 days (week 52).
Time Frame: Baseline (week 0), week 52
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Beats per minute (beats/min)
Arm/Group | Semaglutide | Insulin Aspart
Number analyzed (Participants) | 784 | 765
Beats per minute (beats/min) | 2.2 (8.7) | 1.1 (8.7)

24. Secondary Outcome: Change From Baseline to Week 52 in 36-item Short Form Health Survey Version 2 (SF-36v2): Total Summary Scores (Physical Component and Mental Component) and Scores From the 8 Domains
Description: SF-36v2 is 36-item patient-reported survey of patient health to measure participant's overall health-related quality of life (HRQoL). It has 36 items: 8 domains of physical, mental health status (physical functioning, role physical health (range:21.23-57.16), bodily pain (range: 21.68-62.00), general health (range: 18.95-66.50), vitality (range: 22.89-70.42), social functioning (range: 17.23-57.34), role emotional problem (range: 14.39-56.17) and mental health (range: 11.63-63.95)) and 2 total summary scores: physical components summary (range: 7.32-70.14) and mental components summary (range: 5.79-69.91) calculated from domain scores. All 10 scores range from 5.79-70.42 . Higher scores indicated a better health state. Change from baseline in SF-36v2, 2 summary and 8 domains scores at week 52 is presented. Data is reported for 'on-treatment' observation period: from date of first dose of trial product (week 0) to last date on trial product with a visit window of +7 days (week 52).
Time Frame: Baseline (week 0), week 52
Population: Full analysis set included all randomized participants. Overall Number of Participants Analyzed = participants with available data for this outcome measure and Number Analyzed = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Semaglutide | Insulin Aspart
Number analyzed (Participants) | 803 | 794
Scores on a scale
  Physical Component Summary: number analyzed (Participants) | 802 | 791
  Physical Component Summary | 1.4 (6.4) | 0.4 (6.7)
  Mental Component Summary: number analyzed (Participants) | 802 | 792
  Mental Component Summary | 0.1 (8.6) | -0.3 (8.4)
  Physical Functioning: number analyzed (Participants) | 803 | 793
  Physical Functioning | 1.4 (7.7) | 0.2 (7.8)
  Role Physical Health: number analyzed (Participants) | 802 | 794
  Role Physical Health | 0.1 (7.8) | -0.2 (8.0)
  Bodily Pain: number analyzed (Participants) | 802 | 793
  Bodily Pain | 1.5 (9.0) | 0.8 (9.8)
  General Health | 1.6 (8.0) | 0.3 (8.0)
  Vitality: number analyzed (Participants) | 802 | 792
  Vitality | 1.1 (8.6) | 0.1 (7.9)
  Social Functioning: number analyzed (Participants) | 802 | 793
  Social Functioning | 0.2 (9.5) | -0.6 (9.1)
  Role Emotional Problem: number analyzed (Participants) | 802 | 793
  Role Emotional Problem | 0.0 (9.4) | -0.2 (9.8)
  Mental Health: number analyzed (Participants) | 802 | 792
  Mental Health | 0.6 (8.7) | 0.1 (8.7)

25. Secondary Outcome: Change From Baseline to Week 52 in Diabetes Quality of Life Clinical Trial Questionnaire (DQLCTQ-R): Scores From the 8 Domains
Description: The DQLCTQ-R questionnaire was used to assess participants' HRQoL. The DQLCTQ-R questionnaire contains 57 items and measures and provide scores for the 8 domains (physical function, energy or fatigue, health distress, mental health, satisfaction, treatment satisfaction, treatment flexibility and frequency of symptoms). The 8 domain scores related to DQLCTQ-R are measured on a scale from 0-100. For all scores, higher values indicated better health status. Change from baseline in DQLCTQ-R 8 domain scores at week 52 is presented. Data is reported for 'on-treatment' observation period: from the date of first dose of trial product (week 0) to the last date on trial product with a visit window of +7 days (week 52).
Time Frame: Baseline (week 0), week 52
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Semaglutide | Insulin Aspart
Number analyzed (Participants) | 802 | 795
Scores on a scale
  Physical function: number analyzed (Participants) | 802 | 794
  Physical function | 2.4 (24.6) | -0.4 (26.4)
  Energy or fatigue: number analyzed (Participants) | 802 | 794
  Energy or fatigue | 2.3 (13.0) | 0.4 (12.9)
  Health distress: number analyzed (Participants) | 801 | 794
  Health distress | -0.2 (12.4) | 0.3 (13.2)
  Mental health: number analyzed (Participants) | 800 | 795
  Mental health | 7.2 (18.5) | 0.5 (20.2)
  Satisfaction: number analyzed (Participants) | 799 | 794
  Satisfaction | 4.1 (18.6) | -0.2 (16.2)
  Treatment satisfaction: number analyzed (Participants) | 799 | 792
  Treatment satisfaction | 9.9 (23.9) | 0.8 (24.4)
  Treatment flexibility: number analyzed (Participants) | 798 | 794
  Treatment flexibility | 4.2 (20.1) | -1.2 (19.8)
  Frequency of symptoms: number analyzed (Participants) | 798 | 794
  Frequency of symptoms | 4.1 (15.5) | 1.8 (14.7)

ADVERSE EVENTS:
Time Frame: From week 0 to week 52
Description: All presented adverse events (AEs) are treatment-emergent (i.e., TEAEs). TEAEs were defined as AEs with onset during the 'on-treatment' observation period. Results are based on the safety analysis set (SAS) which included all participants exposed to at least one dose of trial product. One participant died after completing end-of-study visit by an ongoing AE which created discrepancies between all cause mortality deaths and participant flow deaths.
Arm/Group | Semaglutide | Insulin Aspart
All-Cause Mortality (participants affected / at risk) | 12/874 | 1/864
Serious Adverse Events (participants affected / at risk) | 65/874 | 84/864
Other Adverse Events (participants affected / at risk) | 225/874 | 65/864
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide (N=874) | Insulin Aspart (N=864)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abscess sweat gland (Infections and infestations) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 3 (4) | 4 (4)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adhesion (General disorders) | 1 (1) | 0 (0)
Anal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 2 (2)
Angina unstable (Cardiac disorders) | 1 (1) | 1 (1)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1)
Aortic valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 2 (2)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 3 (3)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1)
Bladder perforation (Renal and urinary disorders) | 0 (0) | 1 (1)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bradyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Brain stem infarction (Nervous system disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 3 (3) | 2 (2)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 1 (2)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 3 (3)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 4 (4) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 3 (4)
Death (General disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (2) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic gangrene (Infections and infestations) | 1 (1) | 0 (0)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 0 (0) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Electric shock (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Embolic cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Empyema (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 3 (3) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypoglycaemia unawareness (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemic coma (Nervous system disorders) | 0 (0) | 1 (1)
Hypoglycaemic seizure (Nervous system disorders) | 1 (1) | 0 (0)
Hypoglycaemic unconsciousness (Nervous system disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 1 (1) | 0 (0)
Inflammatory pseudotumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
Intraductal papilloma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 2 (2) | 4 (4)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Macular oedema (Eye disorders) | 0 (0) | 1 (1)
Metastases to gastrointestinal tract (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 3 (4) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Optic ischaemic neuropathy (Eye disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 2 (3)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 1 (2) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 5 (6)
Postoperative wound infection (Infections and infestations) | 2 (2) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Removal of internal fixation (Surgical and medical procedures) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal abscess (Infections and infestations) | 1 (1) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Thalamic infarction (Nervous system disorders) | 0 (0) | 1 (1)
Therapeutic procedure (Surgical and medical procedures) | 0 (0) | 1 (1)
Toe amputation (Surgical and medical procedures) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular stent stenosis (General disorders) | 0 (0) | 1 (1)
Vertebrobasilar insufficiency (Nervous system disorders) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 1 (1)
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Wrong product administered (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide (N=874) | Insulin Aspart (N=864)
Diarrhoea (Gastrointestinal disorders) | 65 (98) | 23 (29)
Nasopharyngitis (Infections and infestations) | 57 (69) | 51 (73)
Nausea (Gastrointestinal disorders) | 129 (174) | 7 (7)
Vomiting (Gastrointestinal disorders) | 50 (78) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2020-07-08): https://cdn.clinicaltrials.gov/large-docs/74/NCT03689374/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-25): https://cdn.clinicaltrials.gov/large-docs/74/NCT03689374/SAP_001.pdf